CLINICAL TRIAL: NCT01896453
Title: Treatment of Chronic Non-specific Low Back Pain With Brain and Peripheral Electrical Stimulation: a Factorial, Randomized Controlled Trial
Brief Title: Brain and Peripheral Electrical Stimulation in Chronic Low Back Pain: a Factorial Design
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: tDCSBACKPAIN; USaoPauloGH (Other: USaoPauloGH)
Record Dates: First submitted 2013-06-19; First posted 2013-07-11 (Estimated); Last update posted 2014-12-04 (Estimated); Status verified 2013-10

CONDITIONS: Chronic Low Back Pain
MeSH Terms: interventions — Transcranial Direct Current Stimulation; Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- tDCS real + TENS real (Active Comparator): Real transcranial direct current stimulation associated with real transcutaneous electrical nerve stimulation (TENS).
  tDCS: 20 minutes, 2mA, primary motor cortex anode (contralateral to the lesion) and supraorbital cathode (ipsilateral to the lesion).
  TENS: 40 minutes, 100Hz, 200µs, 2 channels with electrodes over the low back area of pain.
  Interventions: Procedure: Transcranial direct current stimulation (tDCS); Procedure: Transcutaneous electrical nerve stimulation (TENS)
- tDCS real + TENS sham (Experimental): Real transcranial direct current stimulation associated with sham transcutaneous electrical nerve stimulation (TENS).
  tDCS: 20 minutes, 2mA, primary motor cortex anode (contralateral to the lesion) and supraorbital cathode (ipsilateral to the lesion).
  TENS: 40 minutes (30 seconds ON), 100Hz, 200µs, 2 channels with electrodes over the low back area of pain.
  Interventions: Procedure: Transcranial direct current stimulation (tDCS); Procedure: Transcutaneous electrical nerve stimulation (TENS)
- tDCS sham + TENS real (Experimental): Sham transcranial direct current stimulation associated with real transcutaneous electrical nerve stimulation (TENS).
  tDCS: 20 minutes (30 seconds ON), 2mA, primary motor cortex anode (contralateral to the lesion) and supraorbital cathode (ipsilateral to the lesion).
  TENS: 40 minutes, 100Hz, 200µs, 2 channels with electrodes over the low back area of pain.
  Interventions: Procedure: Transcranial direct current stimulation (tDCS); Procedure: Transcutaneous electrical nerve stimulation (TENS)
- Sham tDCS + Sham TENS (Sham Comparator): Sham transcranial direct current stimulation associated with sham transcutaneous electrical nerve stimulation (TENS).
  tDCS: 20 minutes (30 seconds ON), 2mA, primary motor cortex anode (contralateral to the lesion) and supraorbital cathode (ipsilateral to the lesion).
  TENS: 40 minutes (30 seconds ON), 100Hz, 200µs, 2 channels with electrodes over the low back area of pain.
  Interventions: Procedure: Transcranial direct current stimulation (tDCS); Procedure: Transcutaneous electrical nerve stimulation (TENS)

INTERVENTIONS:
Procedure: Transcranial direct current stimulation (tDCS) — Technique based on the application of weak, direct electrical current to the brain through relatively large electrodes that are placed over the scalp, in which anodal and cathodal stimulation increases and decreases cortical excitability, respectively
Procedure: Transcutaneous electrical nerve stimulation (TENS) — Technique based on the application of low-voltage electrical current to the skin through relatively large electrodes that are placed over the pain area.

SUMMARY:
The purpose of this study is to evaluate the efficacy of brain and peripheral electrical stimulation on chronic non-specific low back pain patients.

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged > 18 years and <65 years
* Complaining of back pain for more than three months
* Presence of a chronic pain measurable with the number rating scale (NRS 0-10) not less than 4 during a 1 week daily NRS monitoring
* Seeking care for low back pain

Exclusion Criteria:

* Previous surgery on the spine, spondylolisthesis
* Previous treatment with TENS <6 months
* Previous treatment with tDCS
* Disc herniation with nerve compression
* Neurological, psychiatric and rheumatologic diseases
* Impaired sensibility
* Use of pacemakers or other implanted devices
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2013-06; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Pain intensity | Four weeks after randomization
  Pain intensity will be evaluated by numerical rating scale (0-10).

SECONDARY OUTCOMES:
Disability | 4 weeks, 3 and 6 months after randomization.
  The Roland Morris disability questionnaire (RMDQ) is composed of 24 yes or no questions designed to assess disability related to back pain.
Quality of pain | 4 weeks, 3 and 6 months after randomization.
  The Short form of the McGill pain questionnaire (SF-MPQ) consists of 15 representative words from the sensory and affective categories of the standard long form. The 6 point intensity scale and a VAS are included to provide indices of overall pain intensity.
Global perceived effect (GPE) | 4 weeks, 3 and 6 months after randomization.
  Global perceived effect is an 11 point scale that ranges from 5 (vastly worse) through 0 (no change) to 5 (completely recovered). For all measures of global perceived effect (at baseline and all follow-ups), participants were asked compared to when this episode ﬁrst started, how would you describe your back these days. A higher score indicates higher recovery from the condition.
Pain intensity | 3 and 6 months after randomization
  Pain intensity will be evaluated by numerical rating scale (0-10)

OTHER OUTCOMES:
Anxiety | 4 weeks, 3 and 6 months after randomization.
  Visual analogue scale (VAS)for anxiety assesses anxiety symptoms that we tracked as possible confounding factor.
Depression | 4 weeks, 3 and 6 months after randomization
  Beck depression inventory (BDI) for depressive symptoms that we tracked as possible confounding factor.
Satisfaction with care | 4 weeks after randomization
  Satisfaction with care will be measured by the Medrisk Instrument for Measuring Patient Satisfaction with Physiotherapy Care.

CONTACTS AND LOCATIONS:
Overall Officials: Fuad A Hazime, PT, Principal Investigator — University of Sao Paulo; Silvia MA João, PT, Study Chair — University of Sao Paulo
Locations (1):
- School of Physiotherapy - University of São Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Hazime FA, de Freitas DG, Monteiro RL, Maretto RL, Carvalho NA, Hasue RH, Joao SM. Analgesic efficacy of cerebral and peripheral electrical stimulation in chronic nonspecific low back pain: a randomized, double-blind, factorial clinical trial. BMC Musculoskelet Disord. 2015 Jan 31;16(1):7. doi: 10.1186/s12891-015-0461-1. PMID 25636503